CLINICAL TRIAL: NCT03210129
Title: Motivational Interviewing to Increase Physical Activity Behaviour in Breast, Endometrial and Colorectal Cancer Patients in the Grand-Duchy of Luxembourg: a Pilot Randomized Controlled Trial
Brief Title: Motivational Interviewing to Increase Physical Activity Behaviour in Cancer Patients
Acronym: MIPAClux
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luxembourg Institute of Health (Other Government)
Collaborators: Fondation Cancer (Unknown)
Responsible Party: Principal Investigator, Laurent Malisoux, PhD, PhD, Luxembourg Institute of Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DoPH_SMRL_20161208
Record Dates: First submitted 2017-06-26; First posted 2017-07-06 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Cancer, Breast; Cancer of Colon; Endometrial Cancer
Keywords: Motivation; Behavior; Exercise; Motivational interview; Cancer; economic evaluation
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Endometrial Neoplasms; Behavior; Motor Activity; Neoplasms | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: The patients will be randomly assigned to the experimental group with motivational interviewing or the control group. Group assignment will be done by a motivational interviewing counsellor using randomization lists generated by the Competence Center in Methodology and Statistics (Luxembourg Institute of Health). For each type of cancer, a separate randomisation list will be used.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Every patient will be given a person-specific code and every information collected will be pseudonymised.
  The group assignment will be hidden to the investigator and to the scientific collaborators who will collect, record and analyse the data. However, both patients and the two motivational interviewing counsellors will be aware of the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational interviewing (Experimental): Patients of the motivational interviewing group will receive standard care alongside motivational interviewing to change their behavior regarding physical activity.
  Interventions: Behavioral: Motivational interviewing
- Control Group (No Intervention): Patients of the control group will receive standard care alone.

INTERVENTIONS:
Behavioral: Motivational interviewing — the patients of the motivational interviewing group will receive 12 motivational interviewing sessions within 12 weeks: 2 face-to-face sessions and 10 phone call sessions. The first and the seventh motivational interviewing sessions will be face-to-face sessions. An intervention is considered valid if a minimum of 10 sessions has been completed. The face-to-face motivational interviewing sessions will be administered at the Luxembourg Institute of Health (Strassen, Luxembourg). They generally last up to 30 minutes, while the motivational interviewing phone calls generally last up to 15 minutes. Thereby, patients in the motivational interviewing group will receive a total of approximately 3.5 hours of contact time over a period of 12 weeks.
  Motivational interviewing techniques will explore self-assessed confidence, ambivalence, and personal values concerning changes in active lifestyle.
  Arms: Motivational interviewing

SUMMARY:
Physical activity is not only efficient for primary prevention of several cancer types, but it also plays an important role in cancer survivors. Physical activity after a cancer diagnosis has been associated with reduced overall and cancer-specific mortality. It has significant positive effects on physical fitness and several cancer-related symptoms including fatigue, sleep disturbance, depression and anxiety. The evidence is considerable and consistent for breast, colorectal and endometrial cancers. However, patients are generally insufficiently active, and participation rates in physical activity opportunities offered by specialized organizations are low. This pilot study will evaluate the feasibility, efficacy and cost-effectiveness of an intervention seeking to increase active lifestyle and physical activity participation of cancer patients. To encourage this behavioural change, motivational interviewing will be used, a patient-centred approach aimed at increasing the patients' motivation for a behavioural change through open-ended discussions.

Seventy patients with breast, colorectal or endometrial cancer will be recruited within a time period of 12 months. Patients will be randomly assigned to an intervention or a control group. The intervention group will receive standard care alongside 12 motivational interviewing sessions within 12 weeks. The control group will receive standard care only. Physical activity behaviour (3D-accelerometer) and physical fitness (cardiovascular and strength fitness) will be measured in the week preceding and following the intervention. Additionally, a subgroup from both study arms will be assessed 12 weeks after the completion of the intervention. The investigators hypothesize that sedentary time will decrease and time spent in moderate and vigorous physical activity, physical fitness and quality of life of cancer survivors will increase to a greater extent in the intervention group than in the control group. Furthermore, health-related quality of life and resource use (intervention and healthcare costs, out of pocket costs) will be measured to evaluate the cost-effectiveness of the intervention.

DETAILED DESCRIPTION:
All recruited patients will receive the same standard care, only those who will be allocated to the experimental group will receive the intervention. This project will run over total period of 21 months. Patients will be offered to join the project over a duration of 12 months. With the help of oncologists and surgeons, an oral agreement will be collected from the eligible patients who agree to be contacted by an investigator of the study. Once the patients have entered the study, they will be followed for 26 weeks, including 12 weeks of intervention or control period and 12 weeks of follow-up to evaluate if the expected intervention-induced behavioural change is maintained:

* Week 1: inclusion and first visit. The patients will be contacted (phone call) by an investigator who will provide explanations about the study. Notably, the investigator will explain that the patients will be allocated randomly to one of two study arms and that they may not chose which one they will be allocated to. In addition, the investigator will check eligibility through a brief questionnaire-based interview. Patients who meet the inclusion criteria will be invited to come to the Luxembourg Institute of Health (Strassen, Luxembourg) for the first visit. During this first visit (duration: 90 min), patients will be asked to sign the written informed consent. Then, patients will be asked to fill in several questionnaires available in English, French, German and Portuguese: three background questionnaires and one cancer-specific health related quality of life (HRQoL) questionnaire (EORTC-QLQ30). Height and weight will be measured. Patients will subsequently perform physical fitness tests, including ramped Bruce protocol test on a treadmill, leg strength and grip strength tests. Finally, patients will receive a 3D-accelerometer (Actigraph) measuring physical activity behaviour, which they will have to wear for one week. Further details one these methodologies are provided below.
* End of week 1: phone call. An investigator will call the patients one day before the end of the recording period of physical activity to remind them to send back the accelerometer. Furthermore, patients will reply by telephone to the generic HRQoL questionnaire (EQ-5D-5L questionnaire, please see details of this questionnaire in the "Cost-effectiveness of the intervention" section). This questionnaire will be administered repetitively throughout and at the end of the intervention.
* Week 2 to week 13: intervention. During a period of 12 weeks, the patients in the intervention group will attend 2 face-to-face and 10 telephone motivation interviewing sessions (please see details in the "Intervention" section). The patients entering the control group will not receive this specific treatment during that period.
* Week 5: phone call. The patients will be called to answer the EQ-5D-5L questionnaire.
* Week 9: phone call. The patients will be called to answer the EQ-5D-5L questionnaire.
* Week 13: phone call. Patients will be called for a reminder of the second visit date (already determined during the first visit).
* Week 14: second visit. Patients will be invited to come to the Luxembourg Institute of Health (Strassen, Luxembourg). During this second visit (duration: 70 min), patient will fill in the EORTC-QLQ30 questionnaire and the cost questionnaire (please see details of this questionnaire in the "Cost-effectiveness of the intervention" section). Height and weight will be measured. Patients will perform the same physical fitness tests as during the first visit (ramped Bruce protocol on a treadmill, leg strength and grip strength). Patients will be handed out the accelerometer to be worn during one week to evaluate their physical activity behaviour.
* End of week 14: phone call. An investigator will call the patients one day before the end of the recording period of physical activity to remind them to send back the accelerometer and to answer the EQ-5D-5L questionnaire.
* Week 14 to week 25: follow-up.
* Week 25: Phone call. Patients will be called for a reminder of the third visit date (already determined during the second visit).
* Week 26: third visit. Patients will be invited to come to the Luxembourg Institute of Health (Strassen, Luxembourg). During this third visit (duration: 70 min), patient will fill in the EORTC-QLQ30 questionnaire and the cost questionnaire. Height and weight will be measured. Patients will perform the same physical fitness tests as during the first and second visits (ramped Bruce protocol on a treadmill, leg strength and grip strength). Patients will be handed out the accelerometer to be worn during one week to evaluate their physical activity behaviour.
* End of week 26: phone call. An investigator will call the patients one day before the end of the recording period of physical activity to remind them to send back the accelerometer and to answer the EQ-5D-5L questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* breast, endometrial or colorectal cancer
* cancer stage ≤ stage III
* > 3 months after primary treatment
* < 24 months after primary treatment
* ECOG performance score < 2
* Signed Informed consent

Exclusion Criteria:

* recurrent cancer
* history of other types of cancer
* second primary tumor
* planned surgery within the duration of the study
* known or obvious cognitive or psychiatric impairments
* positive pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Change in physical activity behavior | week 1, week 14 and week 26
  An objective measurement of the patients' physical activity behaviour will be conducted using the ActiGraph™ GT3X+, a validated 3D-accelerometer, which will be used together with the corresponding ActiLife 6™ data analysis software. Physical activity behaviour will be measured three times (week 1, week 14 and week 26).
  The main outcome is the change between week 1 and week 14.

SECONDARY OUTCOMES:
Body mass index | week 1, week 14 and week 26
  Body mass index will be calculated based on height and weight, combined to report BMI in kg/m^2. Height will be measured with a height gauge. Weight will be measured with a weighing machine.
Ramped Bruce Protocol test | week 1, week 14 and week 26
  patients will start to walk at an initial speed set at 1.6 km/h on the treadmill on a horizontal position. Subsequently, the speed and the slope will be increased progressively according to the stages of a predefined protocol. The outcome will be the exercise stage reached at 85% of the maximal heart rate.
30 seconds chair test | week 1, week 14 and week 26
  Patients will rise to a full standing position and then sit back down again, repeating this movement for 30 seconds. The total number of repetitions will be recorded.
Southampton protocol | week 1, week 14 and week 26
  The best of six grip strength measurements will be used in statistical analyses.
Cost-effectiveness of the intervention | week 1 (quality of life and cost questionnaires), week 4 (quality of life questionnaire), week 8 (quality of life questionnaire) week 14 (quality of life and cost questionnaires) and week 26 (quality of life and cost questionnaires)
  A decision analytic model will be developed to calculate the cost-effectiveness of motivational interviewing based on quality of life and cost questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Malisoux, PhD, Principal Investigator — Luxembourg Institute of Health; Alexis Lion, PhD, Study Director — Luxembourg Institute of Health
Locations (1):
- Luxembourg Institute for Health, Luxembourg, Luxembourg

IPD SHARING:
Plan to Share IPD: No
The IPD will not be shared.

REFERENCES:
- See also: Official website of the Luxembourg Institute of Health — https://www.lih.lu/
- See also: Website of Sport-Santé which provides theoretical and practical information regarding exercise and health — http://www.sport-sante.lu